CLINICAL TRIAL: NCT05554848
Title: Efficacy of Dexmedetomidine and Magnesium Sulfate in Preventing Postoperative Junctional Ectopic Tachycardia After Pediatric Cardiac Surgery: Randomized Controlled Trial
Brief Title: Dexmedetomidine and Magnesium Sulfate in Preventing Junctional Ectopic Tachycardia After Pediatric Cardiac Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Mohamed Elhaddad, Lecturer of Anesthesia, ICU and Pain managment, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: N-62-2022
Record Dates: First submitted 2022-09-19; First posted 2022-09-26 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Post Operative Arrythmia
MeSH Terms: interventions — Dexmedetomidine; Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- control group (No Intervention): patients will receive normal saline instead of dexmedetomidine and MgSo4 .
- dexmedetomidine group (Active Comparator): patients will receive the same of dexmedetomidine as MD group in addition to normal saline instead of Magnesium Sulfate .
  Interventions: Drug: Dexmedetomidine
- Dexmedetomidine Mgso4 group (Active Comparator): patients will receive dexmedetomidine 0.5 µg/kg diluted in 50 mL of normal saline intravenously over 20 minutes, After induction followed by 0.5 µg/kg per hour infusion for 72 hours postoperatively or ready for extubation prior to 72 hour time period (Precedex ; Hospira Worldwide ,Lake Forest, IL).(20) and receiving Magnesium Sulfate (50 mg/kg) bolus administered at the time of Aortic Cross Clamp Release. with continued administration for 72 hours postoperatively at a dose of 30 mg/kg/day
  Interventions: Drug: Dexmedetomidine; Drug: Magnesium sulfate

INTERVENTIONS:
Drug: Dexmedetomidine — dexmedetomidine 0.5 µg/kg diluted in 50 mL of normal saline intravenously over 20 minutes, After induction followed by 0.5 µg/kg per hour infusion for 72 hours postoperatively or ready for extubation prior to 72 hour time period
  Other Names: Precedex
  Arms: Dexmedetomidine Mgso4 group; dexmedetomidine group
Drug: Magnesium sulfate — Magnesium Sulfate (50 mg/kg) bolus administered at the time of Aortic Cross Clamp Release. with continued administration for 72 hours postoperatively at a dose of 30 mg/kg/day.
  Arms: Dexmedetomidine Mgso4 group

SUMMARY:
to study the prophylactic effect of magnesium sulfate , dexmedetomidine or their combination in reduction the incidence of JETS postoperative

DETAILED DESCRIPTION:
Following approval from research and ethics committee, preoperative preparation, and anesthesia inductuion. the baseline heart rate (HR) and blood pressure (BP) will be recorded.

The patients will be divided into three groups according to the type of drug injected.

Group MD (dexmedetomidine Mgso4 group): include (40 ) patients and will receive dexmedetomidine 0.5 µg/kg diluted in 50 mL of normal saline intravenously over 20 minutes, After induction followed by 0.5 µg/kg per hour infusion for 72 hours postoperatively or ready for extubation prior to 72 hour time period (Precedex ; Hospira Worldwide ,Lake Forest, IL).(20) and receiving Magnesium Sulfate (50 mg/kg) bolus administered at the time of Aortic Cross Clamp Release. with continued administration for 72 hours postoperatively at a dose of 30 mg/kg/day.(21) Group D (dexmedetomidine group): include (40 ) patients and will receive the same of dexmedetomidine as MD group in addition to normal saline instead of Magnesium Sulfate .

Group C (control group): include (40 ) patients and will receive normal saline instead of dexmedetomidine and MgSo4 .

after the end of the procedure, inhalational anesthetics will be stopped as well the muscle relaxant. The patient will be transferred to the ICU.

In ICU , the post-operative rhythm was monitored to detect the early incidence of arrythmia

Diagnostic criteria for JET included the following:

* Tachycardia with QRS similar to sinus rhythm QRS
* A ventricular rate more than 170 beats/min
* AV dissociation with or without hemodynamic compromise
* A ventricular rate faster than the atrial rate. (8) Early onset postoperative JET was defined as the presence of JET during the first 72 h postoperatively. Continuous ECG monitoring will be used continuously in the PCCU. Standard 12-lead ECG will be registered in all patients preoperatively and at the time of PCCU admission. When JET was detected on the ECG monitor this will be also documented with a standard ECG strip Patients who developed JET and were hemodynamically unstable were managed with mild hypothermia, reduction in inotropes, magnesium, digoxin, and amiodarone.

ELIGIBILITY:
Inclusion Criteria:

* Age: less than 5 yrs.
* Weight: more than 5 kg .
* Pathology :A-V canal ,VSD ,ASD undergoing corrective surgery with normal sinus rhythm, and stable hemodynamics.

Exclusion Criteria:

* a history of arrhythmias within the last 6 months, current use of antiarrhythmic medication such as amiodarone, digoxin.
* patients with pacemaker or atrioventricular (A-V) block.
* known allergy to dexmedetomidine or magnesium sulfate.
* patients with a history of re-do surgery.

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative JET | for 72 hours postoperatively.
  Incidence of postoperative JET for 72 hours postoperatively.

SECONDARY OUTCOMES:
• Vasoactive - inotropic score | for 72 hours postoperatively.
  Inotropic score = (dopamine × 1) + (dobutamine × 1) + (adrenaline × 100) + (noradrenaline × 100) + (milrinone × 10). Dosages of above drugs were in mcg/kg/min
prognostic indices | for 72 hours postoperatively.
  • time to extubation ( in hours), ICU stay (in days) , and hospital stay (in days)

CONTACTS AND LOCATIONS:
Locations (1):
- Kasralainy Faculty of Medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided